CLINICAL TRIAL: NCT05872373
Title: Snakebite Prevention and First Aid Through Community Engagement in Bangladesh
Brief Title: Snakebite Prevention and First Aid Through Community Engagement
Acronym: SPACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Toxicology Society of Bangladesh (Other)
Collaborators: Centre for Injury Prevention and Research Bangladesh (Other); Ministry of Health & Family Welfare, Bangladesh (Unknown)
Responsible Party: Principal Investigator, Professor Mohammad Abul Faiz, President, Toxicology Society of Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D02550
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Snakebite
Keywords: Snake envenomation; Community engagement; Prevention of snakebite; First aid
MeSH Terms: conditions — Snake Bites | interventions — First Aid

STUDY DESIGN:
Intervention Model Description: This study is a community trial for better community engagement and creating awareness of the first aid management and prevention of snakebites through different IEC materials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Cases are the community people in the study area where interventions will be provided to measure the outcome of the study.
  Interventions: Behavioral: Snakebite prevention and first aid

INTERVENTIONS:
Behavioral: Snakebite prevention and first aid — The study will offer a communication strategy to develop an effective narrative by using a mix-media campaign, where IEC materials would be chiefly localized.

SUMMARY:
This study will be a community trial conducted in two Upazila (sub-district) of Bangladesh- Kalapara, Patuakhali district and Shibganj, Chapainawabganj district. Kalapara upazila will be the intervention area and Shibganj will be the control area. From both the control and intervention areas, 30 community clinics will be randomly selected. Each community clinic serves 6,000 people and consists of 3 'wards'. So, the sample size will be 1,80,000 in the control and intervention areas, respectively. We would first perform formative research and survey to comprehend the burden and the community's perception of managing and preventing snakebite incidents. Data gathered through this assessment will contribute to finalizing our study interventions. The major goals of these interventions are to enhance community involvement and first aid awareness. Community participation will be addressed through 'Uthan Boithok' (courtyard meeting), health education sessions in schools, community clinics, and Upazila Health Complex (UHC) by displaying/using IEC (Information, Education, and Communication) materials (posters, flip charts, leaflets etc.), traditional songs on snakebite prevention and first aid management. Other interventions will include short audiovisual clips and community radio broadcasts, the development of Snakebite Support Groups (SBSG), and speedy referral responses. These interventions will be evaluated through a baseline survey, a midline process evaluation, and an end-line survey. The final assessment process will be completed by comparing the findings of the baseline and end-line surveys as well as by using the hospital surveillance system. Estimated cases per year and the number of patients who attended the hospital for treatment will be the main assessment criteria.

In this trial, the primary outcome, the incidence of snakebite cases, will be modelled using a mixed effects Poisson regression model to obtain incidence rate ratios (IRRs) comparing the intervention to the control group.

Therefore, this proposed project's community participation and health system-building initiatives will also help to build community awareness and quick treatment response in rural communities which in the long run will reduce the morbidity and mortality from snakebite incidence in Bangladesh.

DETAILED DESCRIPTION:
General Objective:

To determine the impact of community engagement/awareness on snakebite prevention and appropriate first aid practices after snakebite in Bangladesh.

Specific Objective:

1. To depict the snakebite scenario in the study areas.
2. To conduct formative research for designing the intervention for the prevention and management of snakebites in rural Bangladesh.
3. To design and strategize the implementation framework for awareness building, community engagement, and developing community based SBSG for prevention and proper management of snakebites in rural Bangladesh.
4. To implement the implementation programme according to the designed strategies.
5. To evaluate the impact of the implementation programme in increasing awareness for the prevention of snakebites and improving the management practice for snakebites.

Methodology

Methodological framework:

This study will be a community trial. The overall research process, interventions and evaluation methods are provided below:

1. Formative research will be performed to better understand the community perception regarding the snakebite prevention and management. Data gathered through this assessment will contribute to intervention design, message development, intervention implementation, monitoring, and evaluation. In this phase, In-depth Interviews (IDI) will be conducted among the healthcare professionals to comprehend the perception of snakebite treatment. There will be Focus Group Discussion (FGD) sessions among the community people, volunteers, and community leaders to understand their level of knowledge about snakebite prevention and first aid management.
2. Finalization of Intervention: After the formative research the development of interventions will be in process. The intervention package will be developed utilizing (a) findings of the baseline survey and formative research, (b) a review of existing literature including recommendations of 'Guidelines for the Management of Snakebites' World Health Organization (WHO) South East Asia Region (SEAR) Office 2016 which was prepared by a team of experts where one of us (MAF, Principal Investigator- PI) was involved; adopted recommendations in the National Guideline for Management of snakebite 2019 and training modules prepared by Non Communicable Disease Control (NCDC), Directorate General of Health Services (DGHS), Government of Bangladesh (GOB) for providing training to the community health workers (in Bengali) and medical doctors (in English). The investigators were involved in the development of the guidelines and the learner's guide by organizing a workshop involving key stakeholders.
3. Implementation of Interventions

   After the finalization of interventions, the next steps would be implementation of the interventions for better community engagement and creating awareness for first aid management. The following work packages will be implemented at the community level:

   Work package 1: IEC material development and demonstration

   The preparation of intervention processes; the information, education, and communication (IEC) materials for creating community awareness will be developed in Bengali through participatory involvement of the relevant stakeholders including program personnel, health managers, health care professionals and the community. The work steps and IEC materials will include the following:

   1.1 Collection of existing IEC materials (if any) on snakebite prevention and first aid 1.2 Identification of IEC materials for snakebite prevention and first aid with methods of delivery to the community through the lens of anthropology 1.3 Development of IEC materials in Bengali 1.3.1 Possible IEC materials: 1.3.1.1 Posters 1.3.1.2 Flip chart 1.3.1.3 Leaflet and pamphlet 1.3.1.4 Video film 1.3.1.5 Radio talk and short radio advertisements (with special note to local community radio) 1.3.1.6 Popular writing 1.3.1.7 Traditional song- as for example 'Boyati', 'Gambira' 1.3.1.8 Laminated picture of common venomous and non-venomous snakes Community engagement through small group discussion (Courtyard Meeting) will be arranged using the relevant IEC materials developed by the health care staff/SBSG working in the intervention area of a community clinic.

   Community engagement through multi-stakeholder involvement centring the community clinic of the intervention area.

   Work package 2: Community engagement through multi-stakeholder involvement centring the community clinic of the intervention area. 2.1 Identification of stakeholders relevant to prevention and providing first aid following snakebite. Relevant stakeholders will be identified for prevention and providing first aid following snakebite.

   2.2 Engagement of stakeholders (community group, two representatives of three community support groups + others including Health Assistant, Assistant Health Inspector, Family Welfare Assistant) for prevention and providing first aid following snakebite at the community level (scene) through community education, thus engaging the community centring on the community clinic (self-organized first aid/primary care for snakebite).

   2.3 Formation of Snakebite Support Group (SBSG): 5-member team, 3 SBSG in each community clinic area one for each ward. The SBSG will arrange the health education session (at least five in each ward, a total of 450 such sessions in the intervention upazila) on prevention and first aid; will arrange a team of three-wheeler vehicle drivers (CNG/battery operated auto rickshaw) with mobile phone number known to the community who volunteer to transport bite victims in case of any snakebite; exact cost of transport through volunteer drivers will be reimbursed; community may also travel by other preferable means of transportation that is quickly available to them (for example ambulance).

   Work package 3: Providing community education utilizing the developed IEC materials 3.1 Conducting 450 'Uthan Boithok' (courtyard meeting) using flip-chart materials to be developed (1.3) on prevention and appropriate first aid, and to show photos of relevant venomous vs. non-venomous snakes occurring in the area. Public health measures will be taken.

   Key topics of 'Uthan Boithok ' will include prevention by promoting the use of - 'cot & bed net', torch-light, boots, cleaning the surroundings and interior of houses, avoiding risky behavior, avoiding poultry keeping in the house; and first aid by knowing the 'Do's and Don'ts' based on current evidence and practicing appropriate first aid measures as well as required skills. 'Uthan Boithok ' will be organized by the SBSGs with the support of community health workers/Multi-purpose Health Volunteers (MPHV) of the area and an action plan to be developed by the Upazila coordinator.

   3.2 Conducting regular (bi-weekly) health education at the community clinic by Community Health Care Provider (CHCP) using the flipchart.

   3.3 Utilization of the developed posters on snakebite prevention and first aid developed.

   3.4 Conducting school/college-based seminars and symposia: at least one in each intervention community clinic area.

   Work package 4: Best practice model establishment: Establishing a best-practice model for the clinical management of snakebites in the UzHC of both control and intervention areas. This is essential for ensuring that snakebite patients coming to the UzHC are managed appropriately in the context.

   4.1 Providing training or retraining to a team of health professionals (doctors, nurses, sub-assistant community medical officers) at selected Upazila Health Complex (UzHC) on the clinical management of snakebites.

   4.2 Arranging essential logistics including supply of antivenom and other drugs needed for the management of snakebite envenoming, from the government sources through coordination with relevant Operational Plans (OPs) 4.3 Providing health education by health care professionals on snakebite prevention and appropriate first aid following snakebite to the snakebite victims, their families and the public attending the UzHC.

   4.4 Providing supportive supervision to the health care professionals of UzHC ('spoke') for managing snakebites through a 24/7 online connection with a dedicated medical college or district hospital ('hub'). The implementation of this activity will involve the participation of a pool of volunteers having specialist knowledge of snakebite management from the 'hub' hospital or elsewhere providing telemedicine support to the UzHC staff.

   4.5 Study of the perceptions of snakebite treatment including anti-venom (AV) delivery among the health care professionals in the UzHC, using IDI/Key informant interview (KII).

   Work Package 5: Community and hospital surveillance of snakebites 5.1 Establishing a community surveillance system for snakebite: to record all the cases of snakebite in humans and domesticated animals (e.g., poultry, cattle, goat, pig [if any], dog, cat) happening in the community through a structured questionnaire and house to house search during the survey. Any case of snakebite occurring in the community will be notified to the CHCP of the community clinic by all (including SBSG, community health workers) for monthly onward transfer of basic snakebite data to UzHC covering age, sex, date, and locality of bite.

   5.2. Hospital Surveillance: Recording all the human cases of snakebite attending the UzHC keeping a 'snakebite register' and replicating this for snakebite cases on domesticated animals seen at the veterinary hospital of the upazila and the district (if any). All patients of snakebite attending the UzHC in intervention areas will be reimbursed for availing the quick transport arranged by the SBSG at the community level. Arrangements will be made for keeping the brought killed snake specimen if brought by the victims or their attendants and for appropriately labeling and preserving them in the facility.
4. Evaluation through community survey: The final process will be evaluation. As the process of evaluation, at least two community survey will be conducted. Baseline survey will be conducted before the implementation of the interventions. Midline survey will be undertaken as process of evaluation. Finally, endline survey will be conducted.

Baseline survey:

To evaluate the impact of implementation program in increasing awareness for prevention of snakebite and improving the management practice for snakebite the community survey will be conducted in both the control and intervention area. In this process, a baseline survey will be started simultaneously with formative research.

Study Design: This baseline study will be cross sectional survey to understand the overall scenario of snakebite prevention and first aid management.

Study Setting: This survey will be conducted in the Shibganj upazila of Chapainawabganj and Kalapara upazila of Patuakhali district. It will be conducted in 30 randomly selected community clinic areas of the intervention upazila in one district and control area will be similar 30 community clinic areas in control upazila in another district.

Study population: The study population will be the community people residing in 3 wards of the catchment areas of community clinics in control and intervention area. An eligible participants for the household survey will be people residing in the study area for more than six months. In case of community survey, the key participant will be considered as the head of the family member. Moreover, if other family members can give relevant information about the victim, they can be invited to join the interview.

Data Collection Instruments for study: The tools will be adopted and translated in Bengali for collecting data from the study site in Bangladesh. The data collection tools will be used in the study will be pretested before field data collection. The tools would provide information on the indicators.

Key parameters during community surveys:

Household: Yes/No information from all households (HHs) from control and intervention areas and details of positive cases only (Yes) will be obtained, for snakebite cases on either humans or domesticated animals.

Key informant

Phone number of the informant:

Day after the incident:

Global positioning system (GPS) coordinates of the location where the bite occurred (or its close vicinity):

Snakebite victim: Human/Domestic animal (name of the animal species)

Age of the victim:

Sex: Male/Female/Third gender

If female: Pregnancy status:

Bite date and time Bite site (on body) Bite scene circumstances Day time/nighttime If the snake was seen Could you identify the offending snake: Yes/No; respondent chooses from a set of photos of representative venomous and non-venomous snakes of the area (2 species of cobra, 3 species of krait, Russell's viper, green pit viper, non-venomous species)

The local name of the snake that caused the bite:

Snake was killed/brought to the hospital

First aid provided:

* Pressure immobilization done if the bite is on limbs: Yes/No
* Tourniquet (ligatures) applied: Yes/No, number, if yes: materials used
* Treatment sought: 'ozha'/directly to UzHC/elsewhere (please specify)
* Time taken from bite time to hospital arrival time (if taken to hospital):
* Travel time from home to hospital:

Key symptoms after the bite:

Outcome: Survived/died (verbal autopsy of any deceased/fatal cases) Any sequelae: please specify Cost of treatment in Bangladeshi 'Taka': Direct cost:... Indirect cost:... How was the treatment cost covered: from savings, loan, sale of material wealth, other (specify)

Key points to be recorded in case the snakebite victim is a domestic animal:

1. Snakebite in animal (species and/or type/breed) is confirmed/probable (case definition 21 will be given)
2. Type of the animal: Cattle, buffalo, goats, sheep, pig, poultry, dog, cat, others
3. Where did the bite happen: (circumstance of bite)
4. Location of bite: owner's house or farm/animal shed/field/pasture
5. The part of the body that was bitten: limb/head-neck area/abdomen/thorax/udder/tail/ unknown.
6. Treatment provided
7. Type of treatment
8. Outcome of the victim
9. Cost of treatment in Taka: Direct cost:... indirect cost:...
10. How was the treatment cost covered: from savings, loan, sale of material wealth, other

Note:

• Confirmed if the event was witnessed, and clinical signs were consistent with snakebite envenomation (e.g., swelling, bleeding, ptosis, hypersalivation, respiratory difficulties, paralysis, or sudden death).

Probable if the event was not witnessed but there was evidence of contact with a snake (animal playing, fighting a snake, a snake found close to the animal) or fang marks were found, and clinical signs were consistent with snakebite envenomation.

Data collection tool: Quantitative data for this project will be collected using Computer-aided personal interviewing (CAPI ). A structured questionnaire will be utilized to conduct household survey. Competent use of these strategies can increase the amount of information needed, improve data quality, and reduce the risk of bias. The above methods of data collection will be adjusted to each of the study's objectives, considering of the possibility of gathering information in the field and the desired indicators.

Recruitment and training of field personnel: Recruitment All the data collection personnel will be recruited following the standard recruitment procedure. They will be recruited by inviting applications and based on maturity, previous working experience, group cohesion, education level and ability to collect data. The minimum educational qualification of field personnel will be at least Bachelor's degree from a recognized university. All field personnel will be initially recruited as trainees. A trainee will be finally appointed to a specific post depending on his/her performance in the training. Trainees with the best performances will be recruited as Supervisors. A greater number of persons than required will be recruited as trainees so that those found not suitable later or those who drop out can be replaced. Moreover, females will be included in the field teams to have easy access to the respondents.

Training: Training of 2 days duration will be organized at the Centre for Injury Prevention and Research, Bangladesh (CIPRB) headquarter (HQ) for all the field staff to be recruited for the survey. The training room will be organized with maintaining social distancing. Training for the Interviewers will include a thorough discussion on the overall methodology and each study question, practice session, and role-playing. They will be oriented on the concept of the project, study objectives, purpose and specified indicators and parameters through this training. The training will cover the issues on interview techniques, the format of questionnaires as well as data collection and record keeping procedure. Issues regarding privacy and confidentiality will also be covered in the training. Interviewers will be instructed not to discuss any of the details of the interviews or any of the personal information obtained through the interviews with other persons or within themselves. A well-experienced panel of trainers will facilitate the training sessions to fulfil the need of administering quality data collection, quality assurance and management. All the key personnel of the study and other senior professionals of the research team will be engaged to impart the training.

Monitoring and evaluation:

Through the baseline survey following indicators will be measured for further evaluation and monitoring:

* Estimated cases of snakebite for the last one year
* Estimated cases of snakebite death for the last one year
* Number (%) of patients going to hospital for treatment.
* Number (%) of patients presenting with tourniquet on admission to the health facilities.
* Number (%) of patients who visited traditional healers
* Number (%) of patients presenting with immobilization on admission to the health facilities.

Midline Survey In the midline survey, after approaching the interventions in community level, household survey will be conducted among the same population and after completion of one year, midline process evaluation will be done to understand the impact of interventions.

End-line Survey All the interventions will be continued until the end of the study. After two years, end-line survey will be conducted among the same population. The effect of the community awareness created will be assessed by comparison of the results of a base-line survey with survey conducted in the community's year 2 of the project and through the hospital surveillance system.

5. Data analysis After the community survey, we will proceed for final data analysis. The following measurable outcomes will be considered: estimated cases per 100,000 per year; the mean time (minutes) to hospital; number of patients coming to hospital for treatment; number (%) of patients presenting with tourniquet on admission to the health facilities; number (%) of patients who visited traditional healers, ('ozha') and the number (%) of patients presenting with immobilization on admission to the health facilities.

The primary outcome, the incidence of snakebite cases, will be modelled using a mixed effects Poisson regression model to obtain incidence rate ratios (IRRs) comparing the intervention to the control group. A hierarchical modelling approach will be employed in order to account for nested clustering i.e., participants will be clustered in villages which are nested in the clinic catchment area where they come from. The 95% confidence intervals for the IRRs will be calculated and reported. A mixed effects Negative Binomial regression model will be fitted if there will be over-dispersion in the mean of these count data. All tests of significance will be performed at a 5% significance level. A detailed Statistical analysis plan will be developed and approved prior to database lock. Analyses will be done in Stata or R or any other appropriate software.

Key parameters to be analyzed Estimated cases per year Mean time to hospital

Number of patients who came to the hospital for treatment:

Number of patients having tourniquets Number of patients who visited traditional healers, ('ozha') Number of patients who arrived with immobilization in place

Risk management The risks associated with this project can be categorized into those at local level and general contextual factors.

Local Level: Non-cooperation- there may arise various risks or uncertainties in the field level implementation of such a survey on socially sensitive issues such as respondents may avoid the team. To overcome such risk, survey teams will introduce themselves in the survey area; local upazila health manager, UHFPO is an investigator; will acknowledge social elites and others.

Non response; Other risks and uncertainties like non-response on the part of respondents which will be dealt with through appropriate approaches as and when required. The common practices are: rapport building with the respondent, taking consent from the respondent, making aware about basic interest areas and survey objectives etc.

General Contextual Factors; Coronavirus Disease (COVID) situation- current COVID if changed may hamper the movement of the staff including data collectors involved in this assignment. Government instruction in this regard will be followed considering the safety of the survey team members.

Problems with the capacity of any of the research team members; The problems with the capacity of any of the research team members will be managed by continuous monitoring and communication.

Dropout of the team members; any of the team members may drop out at any time during the survey. Considering such risk, more than the required number of staff will be trained.

Data Confidentiality; maintaining the confidentiality of the data in this survey will be a high priority. As the data will contain information on humans, safety measures will be employed to ensure data protection and safe handling. The consent form, study tools and any other forms linking participants' personal information will be kept in a place inaccessible to unauthorized persons. Upon the permission of investigators, access to both hard copy and softcopy of data will be made. During the training, a separate session will be taken to maintain data confidentiality and management. Proper documentation and storage of the data, files or protocols relevant to data management will be handled with utmost care. Regular backup of the existing data will be conducted at appropriate intervals. All computers being used in the study will have restricted access to unauthorized persons.

Quality assurance; quality assurance system will be developed. Deputy Programme Managers (DPM), Community Based Health Care (CBHC), & Injury snakebite, DGHS, GOB and local Upazila Health & Family Planning Officer (UHFPO) of the two study upazilas are co-investigators. The community-led awareness meetings in the intervention upazila will be facilitated by locally innovative multi-purpose health volunteers (MHV) of SBSG among the community group and community support group with the support of local Community Clinic (CC) led community health workers and elected local union members and will be monitored by the study team guided by UHFPO. The SBSG will be motivated during community engagement training attended by senior members of the research team including PI. The healthcare team at UzHC will be trained on the management of snakebite through a structured existing training module and will have 24/7 contact with a 'hub' led by an investigator (Assistant Professor of Medicine) for providing advice digitally. PI and other co-investigators will do periodic monitoring visits during the study. Survey data will be collected on a mobile device with proper supervision and periodic real-time monitoring. The Toxicology Society of Bangladesh (TSB) will provide administrative and monitoring support through 2 recruited full-time managers, 1 coordinator and 1 Quality Control Officer (quality control checking of survey data).

Data cleaning will be performed prior to database lock and statistical analyses will be done on clean datasets.

Dissemination of results:

A dissemination meeting will be arranged at the end of the study with the relevant officials and stakeholders in consultation with the Ministry of Health and Family Welfare (MOHFW) (funder). The findings of the study will be published in scientific journals and presented at conferences and may be utilized for future research. The relevant results on prevention and first aid of snakebites will also be communicated widely in Bengali including the study.

Utilization of Results:

The principles of sustainable development goals (SDG) include 'Universal Health Coverage', 'reduction of out-of-pocket expenditure' and 'poverty alleviation. The provision of snakebite prevention, first aid and management close to communities at UzHC directly contribute to achieving SDGs as snakebite mainly affects marginalized, rural poor people and farming communities and their livestock. Snakebite at nighttime in and around poor rural housing and walking in darkness for the natural calls are risks. In addition to the health and poverty-related SDGs, other elements of the SDG like those addressing adequate improved rural housing (SDG 11.1), adequate access to lighting/access to electricity (SDG 7), and elimination of outdoor open defecation (SDG 6.2) are all also linked with the problem of snakebite envenoming and other health issues. Thus, the community engagement and health system strengthening activities of this proposed project will also contribute to achieving targets corresponding to these SDGs. In fact, snakebite envenoming can be regarded as a 'litmus test' for the health system to deliver services through the UzHC, and for developing feasible strategies to optimize services at this level.

ELIGIBILITY:
Inclusion Criteria:

* People living within the study area

Exclusion Criteria:

* People not giving consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
People are knowledgeable about the prevention of snakebite, engaged in proper management of snakebite, communities are empowered to address snakebite in their areas. | 2 years
  The outcome will be measured by the following metrics- reduce the visit to the traditional healer, reduce the use of tourniquets, increase the practice of immobilization after bites, reduce the mean time between bite to hospital, and the mean time from home to the hospital.

SECONDARY OUTCOMES:
A comprehensive integrated snakebite prevention and management program developed | 2 years
  The following metrics will be used to measure the outcome-reduction in total snakebite cases, patients visit directly to the hospital, increase in case reporting, the use of antivenom in local hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Aniruddha Ghose, FCPS, Study Chair — Chittagong Medical College and Hospital
Locations (1):
- Kalapara Upazila and Upazila Health Complex, Patuakhali, Bangladesh